CLINICAL TRIAL: NCT07033533
Title: Allopurinol Interferes With the Pathological Mechanisms of Hepatic Decompensation
Brief Title: Allopurinol and Pathogenesis of Cirrhosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Khadija Ahmed Mhrose Glal, dr, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ALLOU
Record Dates: First submitted 2025-06-14; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Cirrhoses, Liver
MeSH Terms: interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo
- allopurinol (Active Comparator)
  Interventions: Drug: Allopurinol Tablet

INTERVENTIONS:
Drug: Allopurinol Tablet — allopurinol 300
  Arms: allopurinol
Drug: Placebo — placebo tablet
  Arms: placebo

SUMMARY:
Hepatic decompensation is a common healthcare issue

. This study was conducted to investigate how allopurinol can interfere with the pathological mechanisms of HD.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 both sex

Exclusion Criteria:

* active GIT bleeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
biomarkers as zonulin, LPS, MMP-13, MDA | 6 MONTHS

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No